CLINICAL TRIAL: NCT03898245
Title: Effectiveness of Transcranial Direct Current Stimulation for Postoperative Pain in Total Knee Replacement Surgery
Brief Title: Effectiveness of Transcranial Direct Current Stimulation for TKR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, Associate professor, Department of Anesthesiology and Pain medicine, SMG-SNU Boramae Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2018/00/0000.0
Record Dates: First submitted 2019-03-29; First posted 2019-04-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Transcranial Direct Current Stimulation; Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active tDCS (Active Comparator): intervention : Intensity 2mA, 30minues, 7 times (post operation in 30min, in 4hrs, and 1 time a day from POD#1 to POD #7) apply tDCS
  Interventions: Device: apply tDCS
- sham tDCS (Sham Comparator): Intensity 2mA, 8 seconds (but looks same as an intervention 30mins), 7 times (post operation in 30min, in 4hrs, and 1 time a day from POD#1 to POD #7) apply tDCS (sham mode)
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: apply tDCS — Intensity 2mA, 20minues, 4 times (post operation in 30min, in 4hrs, next day morning and next day afternoon) anodal tDCS applied over the left DLPFC cathodal tDCS applied over the right DLPFC
  Arms: active tDCS
Device: Sham tDCS — Intensity 0mA, 40 seconds, 4 times (post operation in 30min, in 4hrs, next day morning and next day afternoon) anodal tDCS applied over the left DLPFC cathodal tDCS applied over the right DLPFC
  Arms: sham tDCS

SUMMARY:
Transcranial direct current stimulation (tDCS) is a technique of noninvasive cortical stimulation allowing significant modification of brain function used. Clinical application of this technique could be helpful for pain, Parkinson's disease, dystonia, cerebral palsy and dementia etc. And tDCS is safe with only mild, transient adverse effects. But there is few studies focused to postoperative states.

The aim of this project is to reveal the effect of tDCS for postoperative pain after total knee replacement surgery,

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have scheduled elective spine surgery.

Exclusion Criteria:

* Who has Cognitive dysfunction before surgery.
* Who already has delirium before surgery.
* Who has pain disorder ( like CRPS)
* Who cannot reveal the one's pain.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-05-10 (Estimated)

PRIMARY OUTCOMES:
VAS score | 1hour, 6hours, 24 hours, 48 hours
  the decrease of pain scale in postop state with Visual Analog Scale.

SECONDARY OUTCOMES:
Incidence of Delirium | postop day 1,3,6
  Incidence of Delirium
Consumption of PCA | 24 hours
  The consumption of opioid.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Young Hwang, MD,phD, Principal Investigator — Seoul Metropolitan Government Seoup National University Boramae Medical Center
Locations (1):
- Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lefaucheur JP. A comprehensive database of published tDCS clinical trials (2005-2016). Neurophysiol Clin. 2016 Dec;46(6):319-398. doi: 10.1016/j.neucli.2016.10.002. Epub 2016 Nov 17. PMID 27865707
- [Background] Borckardt JJ, Romagnuolo J, Reeves ST, Madan A, Frohman H, Beam W, George MS. Feasibility, safety, and effectiveness of transcranial direct current stimulation for decreasing post-ERCP pain: a randomized, sham-controlled, pilot study. Gastrointest Endosc. 2011 Jun;73(6):1158-64. doi: 10.1016/j.gie.2011.01.050. Epub 2011 Apr 5. PMID 21470608
- [Background] Borckardt JJ, Reeves ST, Robinson SM, May JT, Epperson TI, Gunselman RJ, Schutte HD, Demos HA, Madan A, Fredrich S, George MS. Transcranial direct current stimulation (tDCS) reduces postsurgical opioid consumption in total knee arthroplasty (TKA). Clin J Pain. 2013 Nov;29(11):925-8. doi: 10.1097/AJP.0b013e31827e32be. PMID 23370085